CLINICAL TRIAL: NCT04190849
Title: The European Paediatric Non-alcoholic Fatty Liver Disease Registry (EU-PNAFLD): a Prospective, Longitudinal Follow-up of Children With Non-alcoholic Fatty Liver Disease
Brief Title: European Paediatric Non-Alcoholic Fatty Liver Disease Registry (EU-PNAFLD)
Acronym: EU-PNAFLD
Status: Recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: The European Association for the Study of the Liver (Unknown); Children's Liver Disease Foundation (Unknown)
Responsible Party: Principal Investigator, Jake Mann, Hepatology registrar, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A094204; 174534 (Other: Integrated Research Application System)
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-alcoholic Fatty Liver; Non-alcoholic Steatohepatitis
Keywords: Cirrhosis; Liver disease; Hepatocellular carcinoma; Type 2 diabetes; Atherosclerosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Liver Diseases; Carcinoma, Hepatocellular; Diabetes Mellitus, Type 2; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — EDTA blood for DNA extraction from patient (+/- both parents) (Fasting) serum for metabolite profiling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-alcoholic fatty liver disease patients: Children (<18 years) with a diagnosis of NAFLD with radiological demonstration of increased liver fat and exclusion of other causes.

SUMMARY:
The EU-PNAFLD (The European Paediatric NALFD Registry) will be a network composed of European centres involved in the care of children with NAFLD, and will include Hepatologists, Endocrinologists, and Scientists, supported by relevant international specialists. This collaboration will build on existing infrastructure (local databases and bio-repositories) and will align with the adult European NAFLD Registry ("EPoS", Elucidating Pathways of Steatohepatitis study) to allow long-term follow-up supported by translational studies. Through an international, well-characterised large-scale cohort, we hope to: facilitate multi-centre clinical trials; extend our understanding of the key disease mechanisms of NAFLD; and establish the natural history of paediatric NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis made under 18 years of age.
* Diagnosis of NAFLD spectrum disease (simple steatosis (NAFL), steatosis with abnormal transaminases, NASH ± fibrosis or cirrhosis)
* Diagnosis established by:

  * Radiological evidence of hepatic steatosis (e.g. increased hepatic echogenicity on ultrasound), with
  * Exclusion of secondary causes (negative serological liver screen for HBV/HCV, caeruloplasmin >0.20g/L, no history of excess alcohol consumption, no evidence of iron overload, and no clinically significant alpha-1 antitrypsin (A1AT) phenotype (i.e. SZ, ZZ, SS), with or without
  * Histology (>5% steatosis and histology consistent with paediatric NAFLD)

Exclusion Criteria:

* Secondary fatty liver disease (e.g. glycogen storage diseases, Wilson disease, viral hepatitis, drug-related, autoimmune hepatitis, type 1 diabetes mellitus)
* Post-transplant fatty liver
* >20g/day ethanol intake

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with NAFLD who have been diagnosed either invasively (i.e. using liver biopsy) or using some form of imaging (USS, MRI, CT, MRS) plus exclusion of secondary causes using an appropriate panel of bloods. This aims to facilitate recruitment from a representative population of children, not just those from specialist centres who have undergone biopsy.
  'Secondary NAFLD' (i.e. drug-induced, post-transplant) are not eligible. Children with insulin resistance syndromes are not specifically excluded however this is not the primary focus of EU-PNAFLD and other condition-specific registries are in existence.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-11-14 (Actual); Primary Completion 2047-11 (Estimated); Study Completion 2047-11 (Estimated)

PRIMARY OUTCOMES:
Survival | 30-year follow-up
  All-cause survival

SECONDARY OUTCOMES:
Cardiovascular morbidity | 30-year follow-up
  CAD, CVA, PAD
Liver morbidity | 30-year follow-up
  Decompensated liver disease, transplantation, HCC development
Asymptomatic progression of liver disease | 30-year follow-up
  Presence of advanced fibrosis (on biopsy or non-invasive imaging)

CONTACTS AND LOCATIONS:
Overall Officials: David B Savage, Principal Investigator — University of Cambridge
Locations (3):
- Maastricht UMC, Maastricht, Netherlands
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Birmingham Children's Hospital, Birmingham

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with researchers outside of the Registry

REFERENCES:
- [Background] Mann JP, Vreugdenhil A, Socha P, Janczyk W, Baumann U, Rajwal S, Casswall T, Marcus C, van Mourik I, O'Rahilly S, Savage DB, Noble-Jamieson G, Lacaille F, Dabbas M, Dubern B, Kelly DA, Nobili V, Anstee QM. European paediatric non-alcoholic fatty liver disease registry (EU-PNAFLD): Design and rationale. Contemp Clin Trials. 2018 Dec;75:67-71. doi: 10.1016/j.cct.2018.11.003. Epub 2018 Nov 5. PMID 30408605

DOCUMENTS (1):
  • Study Protocol (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT04190849/Prot_000.pdf